CLINICAL TRIAL: NCT03308162
Title: Acceptability and Feasibility of a Multicomponent Group Intervention to Initiate Health Behavior Change: The Kickstart Health Program
Brief Title: The Kickstart Health Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Collaborators: Wayne State University (Other); Blue Cross Blue Shield of Michigan Foundation (Other)
Responsible Party: Principal Investigator, Lackman-Zeman, Lori A, PhD, Principal Investigator, Corewell Health East
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-270
Record Dates: First submitted 2017-10-03; First posted 2017-10-12 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Health Behavior
Keywords: Integrated Behavioral Health Care
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: Within subjects repeated measures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group Intervention (Experimental): Cognitive behavioral experiential group therapy for health behavior change
  Interventions: Behavioral: Cognitive behavioral experiential group therapy

INTERVENTIONS:
Behavioral: Cognitive behavioral experiential group therapy — The Kickstart Health Program is a Cognitive-Behavioral Experiential Therapy (CBET) that is administered via a person-centered group therapy format. Participants receive multiple therapeutic components that include psychoeducation, cognitive behavioral therapy, motivational interviewing, mindfulness, and acceptance and commitment therapy. Participants will also meditate and exercise in the group.
  Other Names: Kickstart Health

SUMMARY:
This study is testing the acceptability and feasibility of an active, experiential group therapy for health behavior change within a medical setting.

DETAILED DESCRIPTION:
The purpose of the current study is to offer a preliminary test of feasibility and acceptability for a group intervention, conducted in a primary care setting, that aims to teach skills that initiate health behavior change. Participants will be recruited from a local family medicine clinic and groups will be held on site at the clinic. Patients will be recruited by their physicians and given a baseline survey of their exercise and nutrition behaviors as well as their overall well being and self efficacy to change their health behaviors. Participants can join the group at any time and attend as many sessions as desired. Groups are held 2 times per month and include worksheets, meditations, and exercise. Patients and their providers will be given 2 follow up surveys after 5 and 13 weeks to assess for acceptability and feasibility of the program, as well as health behavior change. Statistical analyses will include multivariate analyses, descriptive analyses, and frequency data collection.

ELIGIBILITY:
Inclusion Criteria:

* A patient of the Beaumont Family Medicine Center - Troy/Sterling Heights
* Access to a computer or electronic device with an internet browser
* Internet connectivity
* Patient verbally confirms during recruitment phone call that they can independently or with minimal assistance complete online surveys
* English speaking

Exclusion Criteria:

* Individuals who do not have regular access to internet connectivity
* Not approved by their physician to complete the group exercises
* Denies the ability to fill out online surveys with minimal assistance
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Acceptability and feasibility | 5 weeks
  Survey measure of acceptability and feasibility of the novel study in a health care setting
Change in acceptability and feasibility from 5 weeks | 13 weeks
  Survey measure of a change in acceptability and feasibility of the novel study in a health care setting

SECONDARY OUTCOMES:
Personal Medical History Questionnaire | Baseline
  Measure of relevant medical history
Health Specific Self Efficacy Scales | Baseline
  Measure of one's belief that one can engage in health behavior and it is important
Change in health specific self efficacy from baseline | 5-weeks
  Measure of one's belief that one can engage in health behavior and it is important
Change in health specific self efficacy from 5-weeks | 13-weeks
  Measure of one's belief that one can engage in health behavior and it is important
Exercise Beliefs and Benefits Scale (EBBS) | Baseline, 5-, and 13-weeks
  Measure of one's belief that one can engage in exercise and it is important
Change in exercise Beliefs and Benefits Scale (EBBS) from baseline | 5-weeks
  Measure of one's belief that one can engage in exercise and it is important
Change in exercise Beliefs and Benefits Scale (EBBS) from 5-weeks | 13-weeks
  Measure of one's belief that one can engage in exercise and it is important
Short Form 8 (SF-8) | Baseline, 5-, and 13-weeks
  Measure of subjective health
Change in SF-8 from baseline | 5-weeks
  Measure of subjective health
Change in SF-8 from 5 weeks | 13-weeks
  Measure of subjective health
International Physical Activity Questionnaire (IPAQ) | Baseline, 5-, and 13-weeks
  Measure of weekly physical activity
Change in International Physical Activity Questionnaire (IPAQ) from baseline | 5-weeks
  Measure of weekly physical activity
Change in International Physical Activity Questionnaire (IPAQ) from 5-weeks | 13-weeks
  Measure of weekly physical activity
Simple Food Frequency Questionnaire (S-FFQ) | Baseline
  Measure of food consumption across different food groups
Change in Simple Food Frequency Questionnaire (S-FFQ) from baseline | 5-weeks
  Measure of food consumption across different food groups
Change in Simple Food Frequency Questionnaire (S-FFQ) from 5-weeks | 13-weeks
  Measure of food consumption across different food groups
Satisfaction with Life Scale (SWL) | Baseline, 5-, and 13-weeks
  Measure of overall well being
Change in Satisfaction with Life Scale (SWL) from baseline | 5-weeks
  Measure of overall well being
Change in Satisfaction with Life Scale (SWL) from 5-weeks | 13-weeks
  Measure of overall well being
The Group Attitude Scale | 5-weeks
  Measure of group cohesion
Change in The Group Attitude Scale from 5-weeks | 13-weeks
  Measure of group cohesion
Height | Baseline
  Measure of self reported high
Weight | Baseline
  Measure of self reported weight
Change in weight from baseline | 5-weeks
  Measure of self reported weight
Change in weight from 5-weeks | 13-weeks
  Measure of self reported weight
Average daily steps | Baseline
  Measure of self reported average daily steps
Change in average daily steps from baseline | 5-weeks
  Measure of self reported average daily steps
Change in average daily steps from 5-weeks | 13-weeks
  Measure of self reported average daily steps

CONTACTS AND LOCATIONS:
Overall Officials: Lori Lackman-Zeman, PhD, Principal Investigator — Corewell Health East
Locations (1):
- Beaumont Family Medicine, Sterling Heights, Michigan, United States

IPD SHARING:
Plan to Share IPD: No